CLINICAL TRIAL: NCT02757391
Title: Pilot Study of Feasibility and Safety of Personalized Autologous CD8+ T Cell Therapy Plus Anti-PD1 Antibody in Advanced Solid Malignancies
Brief Title: CD8+ T Cell Therapy and Pembrolizumab in Treating Patients With Metastatic Gastrointestinal Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0152; NCI-2016-01058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0152 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Adenocarcinoma; Metastatic Cholangiocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Digestive System Carcinoma; Metastatic Esophageal Carcinoma; Metastatic Gastric Carcinoma; Metastatic Pancreatic Adenocarcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IV Esophageal Cancer AJCC v7; Stage IV Gastric Cancer AJCC v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Cholangiocarcinoma; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Immunotherapy, Adoptive; Adoptive Transfer; aldesleukin; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD8 +T cell therapy, pembrolizumab) (Experimental): Beginning 2 days prior to CD8+ T cell infusion, patients receive cyclophosphamide IV over 30 minutes. Patients undergo CD8+ T cell infusion IV over 2 hours on day 0 and receive aldesleukin SC BID on days 1-14. Beginning on day 1 about 24 hours after CD8+ T cell infusion, patients receive pembrolizumab IV over 30-60 minutes on weeks 3, 6, 12, and 15.
  Interventions: Biological: Adoptive Immunotherapy; Biological: Aldesleukin; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Adoptive Immunotherapy — Undergo CD8 +T cell therapy
  Other Names: ACT; ACT Therapy; Adoptive Cell Immunotherapy; Adoptive Cell Transfer; Adoptive Cell Transfer Immunotherapy; Adoptive Cell Transfer Therapy; adoptive cellular immunotherapy; adoptive cellular therapy; cellular adoptive immunotherapy
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I pilot trial studies the side effects of cluster of differentiation 8 (CD8)+ T cells in treating patients with gastrointestinal tumors that have spread to other places in the body. Tumor cells and blood are used to help create an adoptive T cell therapy, such as CD8+ T cell therapy, that is individually designed for a patient and may help doctors learn more about genetic changes in the tumor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving CD8+ T cell therapy and pembrolizumab may work better in treating patients with gastrointestinal tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of using a personalized adoptive T cell therapy in patients with advanced gastrointestinal malignancies.

SECONDARY OBJECTIVES:

I. Assess the persistence of an immune response after T cell infusion. II. Determine the clinical benefit of adoptive T cell therapy in advanced gastrointestinal cancers.

OUTLINE:

Beginning 2 days prior to CD8+ T cell infusion, patients receive cyclophosphamide intravenously (IV) over 30 minutes. Patients undergo CD8+ T cell infusion IV over 2 hours on day 0 and receive aldesleukin subcutaneously (SC) twice daily (BID) on days 1-14. Beginning on day 1 about 24 hours after CD8+ T cell infusion, patients receive pembrolizumab IV over 30-60 minutes on weeks 3, 6, 12, and 15.

After completion of study treatment, patients are followed up for 24 weeks.

ELIGIBILITY:
Inclusion:

1. Histopathologic documentation of pancreatic adenocarcinoma, colorectal adenocarcinoma, cholangiocarcinoma, esophageal cancer and gastric cancer with radiographic evidence of metastatic disease.
2. Male or female subjects greater than or equal to 18 years of age.
3. ECOG/ Zubrod performance status of 0 or 1.
4. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for at least 8 weeks after pembrolizumab is stopped. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal. Acceptable forms of birth control include condom, diaphragm, hormonal, IUD, or sponge plus spermacide. Abstinence is also an acceptable form of birth control.
5. Men must be willing and able to use an acceptable method of birth control, during and for at least 3 months after completion of the study, if their sexual partners are WOCBP.
6. Willing and able to give informed consent.
7. Adequate vein access: consider PICC or other central line.
8. Patients must have adequate tissue (fresh or frozen) available or planned removal of adequate tissue for analysis. At least 250mg of tumor are needed for peptide elution. There is no specific time limit on how long the tissue can remain frozen prior to use. The tissue will be collected and analyzed under Lab protocol PA15-0176.
9. Patients can have any lines (including zero) of prior therapy to sign consent prior to tissue harvest.
10. Toxicity related to prior therapy must either have returned to </= grade 1, baseline, or been deemed irreversible.
11. ELIGIBILITY FOR TREATMENT: ECOG/Zubrod performance status of 0 to 2.
12. Bi-dimensionally measurable disease by radiographic imaging (CT scan) that represents at least one measurable lesion per RECIST v1.1.
13. At least 4 Weeks must have elapsed since the last chemotherapy, radiotherapy or major surgery.
14. Toxicity related to prior therapy must either have returned to less than or equal to grade 1, baseline, or been deemed irreversible.
15. Subjects must have received at least one line of chemotherapy prior to receiving adoptive T cell therapy and should have exhausted standard of care systemic therapy options. The decision to implement the T cell therapy will be at the discretion of the treating physician. The timing and total exposure to chemotherapy will depend on the tumor type in question (more systemic options for breast cancer; fewer for gastric cancer, for example). Due to the heterogeneity of tumors being treated in this protocol, the discretion of the treating physician in terms of timing of immunotherapy will be critical.

Exclusion:

1. EXCLUSION FOR ENROLLMENT: Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, and carcinoma in situ of the cervix.
2. Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception. Women of childbearing potential with a positive pregnancy test within 3 days prior to entry.
3. Significant cardiovascular abnormalities as defined by any one of the following: 1. Congestive heart failure NYHA classes II-IV. Patients with asymptomatic class I CHF may participate in conjunction with a Cardiology consultation. 2. Clinically significant hypotension. 3. Symptoms of coronary artery disease. 4. Presence of arrhythmias in EKG requiring drug therapy.
4. Active and untreated central nervous system (CNS) metastases (including metastasis identified during screening MRI or contrast CT). Patients with asymptomatic, treated metastases may be eligible if their lesion(s) have demonstrated stability over 2 months.
5. Autoimmune disease: Patients with a history of Inflammatory Bowel Disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. Systemic Lupus Erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the Investigator to be unacceptable.
6. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
7. Inadequate organ function at enrollment defined by: WBC less than or equal to 2000/uL. Hct less than or equal to 24% or Hgb less than or equal to 8 g/dL. ANC less than or equal to 1000. Platelets less than or equal to 75,000. Creatinine greater than or equal to 1.5 x ULN OR creatinine clearance >50 ml/min/1.73m2 for patients with creatinine levels above institutional normal limits. AST/ALT greater than or equal to 2.5 x ULN. Bilirubin greater than or equal to 2.0 x ULN
8. Positive screening tests for HIV, Hep B, and Hep C. If positive results are not indicative of true active or chronic infection, the patient can be treated
9. EXCLUSION CRITERIA FOR TREATMENT: WBC less than or equal to 2000/uL. Hct less than or equal to 24% or Hgb less than or equal to 8 g/dL. ANC less than or equal to 1000. Platelets less than or equal to 75,000. Creatinine greater than or equal to 1.5 x ULN OR creatinine clearance >50 ml/min/1.73m2 for patients with creatinine levels above institutional normal limits. AST/ALT greater than or equal to 2.5 x ULN. Bilirubin greater than or equal to 2.0 x ULN
10. Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception. Women of childbearing potential with a positive pregnancy test within 3 days prior to entry.
11. Steroids are not permitted 3 days prior to T cell infusion and concurrently during therapy.
12. Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any anti-PD-1 dose.
14. After the T cell infusion, patients may not be on any other treatments for their cancer aside from those included in the treatment section of the protocol.
15. Coagulation ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or a PTT is within therapeutic range of intended use of anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity defined as grade 3 or 4 non-hematologic or grade 4 hematologic toxicity per Common Terminology Criteria for Adverse Events version 4.0 | Up to 24 weeks
  Will monitor toxicity of the personalized vaccines in using cohorts of size of 5, starting from the 1st patient using the Bayesian approach of Thall, Simon, Estey.

SECONDARY OUTCOMES:
Persistence of an immune response defined by level of tetramer positive T cell population over time after T cell infusion | Up to 24 weeks
Persistence of an immune response defined by T cell interferon gamma release in response to selected personalized peptide antigens | Up to 24 weeks
Persistence of an immune response defined by levels of intracellular cytokine staining of T cells in response to stimulation with personalized peptide antigens | Up to 24 weeks
Persistence of an immune response defined by detection of antigen spreading | Up to 24 weeks
Proportion of patients who have received T cell infusion that is alive and progression free (complete response [CR] + partial response [PR] + stable disease) defined based on response criteria according to Response Evaluation Criteria in Solid Tumors 1.1 | At 12 weeks post infusion
Time to progression | Up to 24 weeks
Response rate (CR + PR) | Up to 24 weeks
  The response rate will be evaluated using a Simon optimal two-stage design.
Overall survival | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org